CLINICAL TRIAL: NCT07314255
Title: The Role of Trop2 in Radioactive Iodine-131 Therapy Sensitivity in Papillary Thyroid Carcinoma
Acronym: ZL2025
Status: Active, not recruiting | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Collaborators: Lin Zhou (Unknown); Zhijun Chen (Unknown); Yu Su (Unknown); Jingxiu Zhong (Unknown); Tianzhu Lu (Unknown)
Responsible Party: Sponsor
Other Study IDs: Trop2 and PTC; 202211013 (Other Grant/Funding Number: Jiangxi Provincial Health Commission)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: PTC; I-131; Trop2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Postoperative paraffin-embedded specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RAI responder: The ¹³¹I treatment-responsive group was defined as patients who achieved successful radioactive iodine therapy (i.e., lesions disappeared or showed no long-term progression after radioiodine uptake).
  Interventions: Radiation: radioiodine-131 therapy
- RAI nonresponder: The ¹³¹I treatment-resistant group was defined as patients meeting any of the following criteria:
  No radioiodine uptake in metastatic tissues during the first ¹³¹I treatment, with insignificant decrease or an increase in serum Tg levels before and after therapy; Partial lesions exhibit radioiodine uptake while others showed no uptaking; Progressive metastatic disease despite evident radioiodine uptake.
  Interventions: Radiation: radioiodine-131 therapy

INTERVENTIONS:
Radiation: radioiodine-131 therapy — surgery, tsh inhibition therapy

SUMMARY:
Clinincal data and pathological specimens from patients who had undergone at least one radioactive iodine-131 (^131I) therapy in the Department of Nuclear Medicine at Jiangxi Cancer Hospital over the past 8-10 years were retrospectively collected (approximately 30-50 cases each in the ^131I treatment-responsive group vs. the ^131I treatment-resistant group). Patients in the ^131I treatment-resistant group underwent ^18F-Trop2 PET-CT imaging.

Inclusion criteria:

1. History of total thyroidectomy with postoperative pathology confirming papillary thyroid carcinoma (PTC);
2. At least one course of ^131I internal radiotherapy.

Exclusion criteria:

1. Presence of other severe comorbidities;
2. Incomplete clinical or follow-up data. The clinicopathological characteristics and Trop2 expression levels in tissue samples were compared between the ^131I treatment-responsive group and the ^131I treatment-resistant group.

Within the ^131I treatment-resistant group, comparisons were made between the rapidly progressing subgroup and the stable-disease subgroup under TSH-suppressive therapy in terms of clinicopathological features, tissue Trop2 expression levels, and SUVmax of metastatic lesions on ^18F-Trop2 PET-CT imaging. Factors influencing progression-free survival and overall survival in ^131I-resistant patients were analyzed.

ELIGIBILITY:
Inclusion Criteria:( 1) History of total thyroidectomy with postoperative pathology confirming papillary thyroid carcinoma (PTC); (2) At least one course of ^131I internal radiotherapy. Exclusion Criteria:(1) Presence of other severe comorbidities; (2) Incomplete clinical or follow-up data.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who had undergone total thyroidectomy with postoperative pathology confirming papillary thyroid carcinoma and at least one radioactive iodine-131 (^131I) therapy in the Department of Nuclear Medicine at Jiangxi Cancer Hospital over the past 8-10 years were retrospectively collected
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-06-10 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Tumor size; | 6-60 months
  Lesion size was determined using CT imaging. Lymph nodes were assessed based on their shortest diameter, while other target lesions were evaluated based on their longest diameter. Each measurable lesion underwent an average measurement derived from a minimum of three readings, with all measurements conducted by the same individual to minimize measurement discrepancies. Response Evaluation Criteria in Solid Tumors (RECIST 1.1) were used to assess treatment response

SECONDARY OUTCOMES:
Serological assessment | 1-60months
  Including serum thyroglobulin (Tg) and serum anti-thyroglobulin antibody levels (TgAb) in thyrotropin-inhibited states, as well as tumor markers such as CEA

CONTACTS AND LOCATIONS:
Overall Officials: lin zhou, Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided
We will share our plan after our results be published